CLINICAL TRIAL: NCT02750241
Title: Pink Warrior-Support Group Toolkit for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-0040
Record Dates: First submitted 2016-04-18; First posted 2016-04-25 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer; Physical Activity
Keywords: active video game; mHealth; cancer survivor; women's health; breast cancer; physical activity; support group; survivorship
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active video game-based intervention (Experimental): This arm will receive the active video game-based intervention, which will include attending 12 weekly group sessions at the UTMB Breast Health Clinic, participate in self-paced home session, and monitor daily, weekly, and monthly steps using Wii Fit Meter. All participant will be provided a water bottle and a tote bag as a token of appreciation for participation.
  Interventions: Behavioral: Active video game-based intervention
- Pedometer (Active Comparator): This arm will receive the pedometer intervention, which will include attending 3 monthly UTMB Breast Cancer Support Group sessions, and monitor daily, weekly, and monthly steps using a pedometer (Digit-Walker CW-700/701). All participant will be provided a water bottle and a tote bag as a token of appreciation for participation.
  Interventions: Behavioral: Pedometer

INTERVENTIONS:
Behavioral: Active video game-based intervention — * Attend 12 weekly group session at the UTMB Breast Health Clinic to play the active video games using Wii Fit U or Xbox 360.
  * Participate in self-paced home sessions
  * Monitor daily, weekly, and monthly steps using Wii Fit Meter
  * Feedback on physical activity and physical function
  Arms: Active video game-based intervention
Behavioral: Pedometer — * Attend 3 monthly UTMB Breast Cancer Support Group Sessions
  * Monitor daily, weekly, and monthly steps using a pedometer (Digi-walker CW-700/701)
  * Feedback on physical activity and physical function
  Arms: Pedometer

SUMMARY:
Breast cancer survivors, from diagnosis until the end of life, go through many transitions. One major transition is the significant decrease of physical activity immediately after diagnosis. Despite the known benefits of physical activity-speeding recovery time and reduced cancer recurrence risk-only 1 in 3 survivors met physical activity recommendations of 150 minutes of moderate-intensity activity per week. Physical activity interventions have shown effectiveness in helping breast cancer survivors increase physical activity during treatment, but limited evidence-based physical activity interventions have been incorporated into the clinic and community. To address this limitation, the investigators are partnering with the UTMB breast cancer support group to conduct a 12-week physical activity intervention, Pink Warrior.

The goal of this study is to compare an intervention that uses active games versus an intervention uses pedometer to encourage physical activity such as walking within breast cancer survivors in active cancer treatment. The study will include breast cancer survivor between the ages of 18 - 70 whom currently gets less than 150 minutes of planned physical activity per week and received a breast cancer diagnosis within 0 to 6 months. Participants will be randomized to participate in the support group using the active video game-based physical activity intervention (Wii and Xbox active games) or to participate in the existing UTMB breast cancer support group with pedometers (Digi-Walker CW-700/701). The investigators hypothesize that by engaging in active video gaming, breast cancer survivors will be motivated to initiate and maintain physical activity during treatment. This will ultimately increase functional capacity and prevent functional disability in breast cancer survivors.

DETAILED DESCRIPTION:
Increasing and maintaining physical activity among female breast cancer (BC) survivors during treatment remains an unresolved problem in BC survivorship care. BC survivors, from diagnosis until the end of life, go through many transitions. One major transition is the significant decline of physical activity immediately after diagnosis. Despite the known benefits of physical activity-speeding recovery time and reduced cancer recurrence risk-less than 30% of survivors met physical activity recommendations. Physical activity interventions have shown effectiveness in helping BC survivors increase activity during treatment, but limited evidence-based activity interventions have been disseminated into the clinic and community. To address this limitation, we are partnering with the UTMB breast cancer support group to conduct a 12-week physical activity intervention, Pink Warrior, which will investigate the feasibility of implementing active video game-based physical activity intervention among BC survivors undergoing treatment within the support group setting. Participants (N = 60) will be randomized to participate in the support group using the active video game-based physical activity intervention or to participate in the existing UTMB breast cancer support group with pedometers. Our specific aims are:

Aim 1: Evaluate the feasibility and acceptability of active video game-based physical activity intervention among BC survivors undergoing treatment within the support group setting. Measures of feasibility will include weekly attendance records, number of completed home-based worksheets, number of participants completing the program activities, technological issues, and adverse events.

Aim 2: Compare the support group using the active video game-based physical activity intervention to the existing UTMB breast cancer support group with pedometer. Primary outcomes will be changes in physical activity. Secondary outcomes will be changes in physical function, dietary pattern, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent
2. Diagnosed with primary female breast cancer within 0 to 6 months period of time
3. English-speaking between the ages of 18 and 70
4. Able to read and write in English
5. Obtained approval from oncologists for the participant to be involved in the physical activity based support group
6. Able to travel to the UTMB Breast Health Center
7. Able to move arms and legs as well as ambulate
8. Able to see TV screen from a distance of 2 to 4 feet

Exclusion Criteria:

1. Being pregnant
2. Dementia
3. Currently engage in ≥150 minutes of planned moderate physical activity per week for the prior week
4. Are involved in another physical activity intervention

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity steps per day as measured by an Actigraph monitor | Change in steps per day from baseline to 14 weeks
  Change in steps per day between 14 weeks and baseline as measured by an Actigraph monitor
Change in physical activity minutes as measured by an Actigraph monitor | Change in physical activity minutes from baseline to 14 weeks
  Change in physical activity minutes between 14 weeks and baseline as measured by an Actigraph monitor

SECONDARY OUTCOMES:
Change in physical function as measured by the Short Physical Performance Battery (SPPB) | Change in physical function from baseline and 14 weeks
  The SPPB consists of six components: repeated chair sit and stands, balance test, semi-tandem stand, tandem stand, side-by-side stand, and eight feet walk
Change in dietary pattern as measured by the Dietary Screener Questionnaire | Change in dietary pattern from baseline and 14 weeks
  Change in dietary pattern from baseline and 14 weeks] [Safety Issue: No] The Dietary Screener Questionnaire used in the National Health and Nutrition Examination Survey 2009-10. The screener captures frequency of fruits, vegetables, dairy/calcium, added sugar, whole grains/fiber, red meat, and processed meat consumption within the past 30 days
Change in quality of life as measured by the Functional Assessment of Cancer Therapy-Breast measure | Change in quality of life from baseline and 14 weeks
  Changes in physical, social, emotional, functional, and additional well-being between 14 weeks and baseline as measured by FACT-B
Change in hand grip strength as measured by hand dynamometer | Change in hand grip strength from baseline to 14 weeks
  Hand dynamometer estimates the muscle strength generated from flexor muscles of the hand and the forearm

OTHER OUTCOMES:
Change in weight | Change in weight from baseline to 14 weeks
  Change in body weight between 14 weeks and baseline as measured by a weight scale in the clinic
Change in waist circumference | Change in waist circumference from baseline to 14 weeks
  Change in waist circumference between 14 weeks and baseline as measured by Seca-203
Change in physical activity minutes, measured by the Community Healthy Activities Model Program for Seniors | Change in physical activity minutes from baseline to 14 weeks
  Self-reported physical activity questionnaire
Change in physical function, measured by PROMIS measure specific to cancer survivors | Change in physical function from baseline to 14 weeks
  Changes in overall self-reported physical functions between 14 weeks and baseline as measured by PROMIS-Ca Bank v1.1-Physical Function
Change in fatigue, measured by PROMIS measure specific to cancer survivors | Change in fatigue from baseline to 14 weeks
  Changes in overall self-reported fatigue level between 14 weeks and baseline as measured by PROMIS-Ca Bank v1.1-Fatigue
Change in exercise motivation, measured by autonomous motivation specific to physical activity | Change in motivation from baseline to 14 weeks
  Behavioral regulation in Exercise Questionnaire-2 will be used
Change in psychological feelings, measured by Psychological Need Satisfaction in Exercise Scale | Change in psychological feelings from baseline to 14 weeks
  Sub-scales included perceived competence, perceived autonomy, and perceived relatedness
Change in self-regulation, measured by Rovinak et al. scale | Change in self-regulation from baseline to 14 weeks
  Sub-scales include exercise goals and exercise plans
Feasibility-Adherence | 14 weeks
  Adherence will be measured by number of participants who completed at least 80% of the program activities.
Feasibility-Attrition | 14 weeks
  Attrition will be measured by percentage of people who dropped out of the intervention program.
Feasibility-Technological Issues | 14 weeks
  Technological issues will be measured by counting number of occurrence
Feasibility-Adverse Events | 14 weeks
  Adverse events will be measured by counting number of occurrence
Acceptability | 14 weeks
  Participant acceptability and satisfaction will be assessed by a questionnaire with 5-point scale responses

CONTACTS AND LOCATIONS:
Overall Officials: Maria Swartz, PhD, MPH, Principal Investigator — The University of Texas Medical Branch
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swartz MC, Lewis ZH, Deer RR, Stahl AL, Swartz MD, Christopherson U, Basen-Engquist K, Wells SJ, Silva HC, Lyons EJ. Feasibility and Acceptability of an Active Video Game-Based Physical Activity Support Group (Pink Warrior) for Survivors of Breast Cancer: Randomized Controlled Pilot Trial. JMIR Cancer. 2022 Aug 22;8(3):e36889. doi: 10.2196/36889. PMID 35994321